CLINICAL TRIAL: NCT05027477
Title: Customized Ablation of the Prostate With the TULSA Procedure Against Radical Prostatectomy Treatment: a Randomized Controlled Trial for Localized Prostate Cancer (CAPTAIN)
Brief Title: A Comparison of TULSA Procedure vs. Radical Prostatectomy in Participants With Localized Prostate Cancer
Acronym: CAPTAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Profound Medical Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCP-10296
Record Dates: First submitted 2021-08-18; First posted 2021-08-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate ablation; high intensity transurethral ultrasound ablation; MRI-guided; minimally invasive; real-time temperature feedback control; prostate cancer; TULSA; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Radical Prostatectomy (Active Comparator): Patients in this group will undergo Radical prostatectomy. There will be about 67 people in this group.
  Interventions: Device: Radical Prostatectomy
- TULSA Procedure (Experimental): Patients in this group will undergo TULSA Procedure. There will be about 134 people in this group.
  Interventions: Device: TULSA Procedure

INTERVENTIONS:
Device: Radical Prostatectomy — If you are in this group, you will get the standard of care treatment used to treat this type of cancer: radical prostatectomy. You will undergo this procedure as per standard clinical practice. A radical prostatectomy is a surgical procedure that removes the prostate gland. This is done by making a surgical incision and removing the prostate gland.
  Arms: Radical Prostatectomy
Device: TULSA Procedure — If you are in this group, you will get the TULSA Procedure. The TULSA Procedure is a minimally invasive procedure that uses directional ultrasound to produce very high temperature to ablate (destroy) targeted prostate tissue. The procedure is performed in a MRI suite (the physician can see the prostate at all times throughout the procedure) and uses the TULSA-PRO system to ablate prostate tissue. The procedure combines real-time MRI with robotically-driven directional thermal ultrasound to deliver predictable, physician-prescribed ablation of the prostate. Minimally invasive here means that the procedure is performed through natural openings in your body (the urethra) instead of creating larger openings like in traditional surgery.
  Other Names: TULSA-PRO
  Arms: TULSA Procedure

SUMMARY:
Men with localized, intermediate risk prostate cancer will be randomized to undergo either radical prostatectomy or the TULSA procedure, with a follow-up of 10 years in this multi-centered randomized control trial. This study will determine whether the TULSA procedure is as effective and more safe compared to radical prostatectomy.

DETAILED DESCRIPTION:
The typical standard of care for patients with localized, intermediate risk prostate cancer is radical prostatectomy, which involves the surgical removal of the prostate. Although radical prostatectomy is effective in terms of controlling the cancer, it may leave men with significant long-term effects in urinary, sexual function like erectile dysfunction and/or incontinence (loss of bladder control), thus reducing quality of life. Preservation of continence (ability to control your bladder) and potency (ability to achieve erection and/or ejaculation) may be significant concerns for men.

Targeted ablation of localized prostate cancer using MRI-guided technology is becoming a favorable option for many men who wish to have their cancer treated but do not wish to compromise their urinary and sexual functions. The TULSA Procedure is a new, minimally-invasive technique that uses real-time MRI-guided technology to guide the delivery of high-energy ultrasound to precisely, and in a customized fashion specific to you, heat and kill the prostate cancer tissue while protecting important surrounding body parts that are important for preserving urinary and sexual function. Minimally invasive here means that the procedure is performed through natural openings in your body (the urethra) instead of creating larger openings like traditional surgery or minimally invasive surgery.

The purpose of this research study is to:

* Test whether the TULSA Study Procedure preserves or improves your quality of life (urinary, bowel and sexual functions) at 12 months post-study treatment compared to standard of care (radical prostatectomy).
* Test how many subjects who undergo the TULSA Study Procedure are free from treatment failure by 3 years post-study treatment compared to subjects who undergo the standard of care (radical prostatectomy). Treatment failure is defined as undergoing other additional prostate cancer treatments, spreading of cancer or death caused by cancer.

About 201 subjects will participate in this study with 67 randomly assigned to the radical prostatectomy group and 134 randomly assigned to the TULSA procedure group. Patients will have a 1 in 3 chance of being assigned to the radical prostatectomy group and a 2 in 3 chance of being assigned to the TULSA group. Following treatment, patients will be followed up for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 40 to 80 years, with >10 years life expectancy
* NCCN (favorable and unfavourable) intermediate-risk prostate cancer on biopsy acquired within last 12 months
* Stage ≤cT2c, N0, M0
* ISUP Grade Group 2 or 3 disease on TRUS-guided biopsy or in-bore biopsy
* PSA ≤20ng/mL within last 3 months
* Treatment-naïve
* Planned ablation volume is < 3 cm axial radius from urethra on mpMRI acquired within last 6 months

Exclusion Criteria:

* Inability to undergo MRI or general anesthesia
* Suspected tumor is > 30 mm from the prostatic urethra
* Prostate calcifications > 3 mm in maximum extent obstructing ablation of tumor
* Unresolved urinary tract infection or prostatitis
* History of proctitis, bladder stones, hematuria, history of acute urinary retention, severe neurogenic bladder
* Artificial urinary sphincter, penile implant, or intraprostatic implant
* Patients who are otherwise not deemed candidates for radical prostatectomy
* Inability or unwillingness to provide informed consent
* History of anal or rectal fibrosis or stenosis, or urethral stenosis, or other abnormality challenging insertion of devices

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2036-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint - proportion of patients who maintain both urinary continence and erectile potency | 12 months post-treatment
  Compare preservation of urinary continence and erectile potency, between the 2 arms. Urinary continence is defined as 'pad-free' (0 pads/day) (per EPIC question 5) and erectile potency is defined as erection firmness sufficient for penetration (per IIEF question 2).
Efficacy endpoint - proportion of patients free from treatment failure | 36 months post-treatment
  Compare the proportion of patients experiencing treatment failure, between the 2 arms. Treatment failure is defined as delivery of any additional intervention for prostate cancer (local or systemic, including adjuvant therapy), or metastatic disease, or prostate cancer-specific death.

SECONDARY OUTCOMES:
Biochemical failure endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare the proportion of patients with biochemical failure between the two arms. Biochemical failure is defined as PSA≥ 0.2 ng/mL for the RP arm or PSA nadir plus 2 ng/mL for the TULSA arm (adapted from Phoenix criteria).
Histological failure endpoint | At 12 month post treatment, and also at 24 months post treatment for patients who undergo a repeat TULSA
  Compare the proportion of patients who have clinically significant disease (defined as ISUP Grade Group 2 or higher) between the two arms.
mpMRI endpoint (for Tulsa arm only) | At 12 month post treatment, and also at 24 months post treatment for patients who undergo a repeat TULSA
  Characterize the effect of the TULSA Procedure ablation on diagnostic multi-parametric MRI, determined using PI-RADS V2 score, compared to baseline.
Salvage-free survival endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare the proportion of patients who are salvage free, between the two arms. Salvage-free survival is defined as freedom from any salvage treatments after the assigned treatment, for both RP arm and TULSA arm. 1 repeat TULSA does not count as Salvage.
Metastases-free survival endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare the proportion of patients who are free from metastatic disease between the 2 arms, based on imaging.
Prostate cancer-specific survival endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare the proportion of patients who die of prostate cancer between the 2 arms.
Overall survival endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare the proportion of patients who die of any cause, between the 2 arms.
Surgical complications endpoint | At the following study visits post treatment: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5 years
  Compare the frequency and severity of all adverse events between the 2 arms, evaluated by attribution and reported in accordance with Clavien-Dindo classification.
Penile rehabilitation endpoint | At the following study visits post treatment: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5 years
  Compare the proportion of patients who undergo penile rehabilitation between the 2 arms (penile rehab includes implant insertion, medication/injection, traction or pump device).
Penile length endpoint | At 1 month and 12 months post-treatment
  Compare the change in penile length from baseline to after treatment, between the 2 arms, as measured by the study doctor.
Blood loss endpoint | During the procedure and immediately after the procedure
  Compare the volume of blood lost between the two arms during treatment.
Transfusion volume endpoint | During the procedure and immediately after the procedure
  Compare the volume of transfused blood between the two arms during treatment.
Inpatient hospital stay endpoint | Immediately after the procedure
  Compare the length of inpatient stay between the two arms.
IIEF-15 Endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare International Index of Erectile Function (IIEF-15) scores (for domains of sexual function) between the two arms at follow up, referenced to baseline. Low scores indicate a worse outcome.
IPSS Endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare International Prostate Symptom Score (IPSS) scores (for urinary function), between the two arms at follow up, referenced to baseline. Minimum score=0, Maximum score=35. Higher scores indicate a worse outcome.
EPIC Endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24 month, and 3, 4, 5, 6, 7, 8, 9, 10 years
  Compare (Expanded Prostate Cancer Index Composite) EPIC scores (for domains of urinary, sexual, bowel, and hormonal function), scored from 0 (worst) to 100 (best) between the two arms at follow up, referenced to baseline.
NRS Endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24, and 36 months.
  Compare Numerical Rating Scale (NRS) ratings (which measures pain intensity), between the two arms at follow up, referenced to baseline. 0 indicates no pain and 10 indicates worst possible pain.
EQ-5D-5L Endpoint | At each visit post treatment throughout the total study follow up: 1, 3, 6, 9, 12, 18, 24, and 36 months.
  Compare the EQ-5D-5L scores (which measures quality of life), between the two arms at follow up, referenced to baseline. Responses are coded as single-digit numbers expressing the severity level selected in each dimension (Mobility, self-care, usual activities, pain/discomfort and anxiety expression), where level 1 indicates no problem and level 5 indicates extreme problem.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (19):
  - Arizona State Urological Institute, Chandler, Arizona
  - East Valley Urological Center, Mesa, Arizona
  - Investigate MD, Scottsdale, Arizona
  - Atlantic Urology Medical Group, Long Beach, California
  - Urology Group of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Comprehensive Urology Medical Group, Los Angeles, California
  - Alarcon Urology Center, Montebello, California
  - Pasadena Urological Medical Group, Pasadena, California
  - Stanford Cancer Center, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The Urology Place, San Antonio, Texas
- Canada (2):
  - Lawson Health Research Institute, London Health Sciences Centre, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
- Turku University Hospital/TYKS, Turku, Southwest Finland, Finland